## **Cover Page:**

**Study Title:** Prognostic Relevance of Fatty Liver Disease for Patients with Chronic Hepatitis B

**Short Title:** Steatohepatitis in Chronic Hepatitis B

Date: December 31st, 2021.

**NCT number:** not available.

## **Study Protocol:**

Project title: Prognostic Relevance of Fatty Liver Disease for Patients with Chronic Hepatitis B

**Project summary:** Fatty liver disease is increasingly recognized in patients with chronic hepatitis B (CHB). Whether concurrent fatty liver disease affects the long-term outcomes of CHB is unclear. The investigators will perform a longitudinal study to investigate the prognostic relevance of concurrent fatty liver disease for patients with CHB receiving antiviral therapy.

## **Project description:**

Rationale: Fatty liver disease has become more prevalent in individuals with CHB, owing to the obesity epidemic. The coexistence of CHB and fatty liver disease, particularly the histologic phenotype of steatohepatitis, can augment liver damage and increase the risk of liver fibrosis. However, there are limited data on the impact of fatty liver disease on clinical outcomes (e.g., cirrhotic complications, hepatocellular carcinoma, need for liver transplantation, and all-cause death) during comprehensive treatment for CHB.

**Objectives:** To determine the long-term effect of concurrent fatty liver disease, particularly a histologic phenotype of steatohepatitis on all-cause mortality and liver-related complications in patients with CHB receiving antiviral therapy at the Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand.

**Methodology:** Retrospective analysis of a prospectively collected database of 408 patients with chronic HBV infection who underwent a liver biopsy for therapeutic decision in initiating antiviral therapy between 2002 and 2008 at Siriraj Hospital, Bangkok, Thailand.

**Data management and analysis:** Prospectively generated liver database that collates clinical, biochemical, and pathological data regarding chronic HBV infection and fatty liver disease. In addition, associated serological results, radiological reports, and patient follow-up/outcomes will

be also reported. Variables will be documented from the date of liver biopsy until either the study

outcomes (death, liver transplantation, or liver-related complications), loss of follow-up, or the

end of the study period.

Statistical analyses will be done using SPSS version 18.0. Quantitative variables will be compared

between groups using standard parametric or non-parametric tests, and qualitative variables will

be compared using the Chi-squared test. The cumulative probabilities of mortality or liver

transplantation and liver-related complications will be estimated by the Kaplan-Meier method

and compared by the log-rank test. Hazard ratios and 95% confidence interval estimates for the

outcomes will be calculated by Cox proportional hazard models.

Ethical considerations: This study is approved by the Institutional Review Board and is conducted

in accordance with the Declaration of Helsinki.

**Gender issues:** None

References

1. Schweitzer A, Horn J, Mikolajczyk RT, et al. Estimations of worldwide prevalence of

chronic hepatitis B virus infection: a systematic review of data published between 1965

and 2013. Lancet 2015;386(10003):1546-1555.

2. European Association for the Study of the L. EASL 2017 Clinical Practice Guidelines on the

management of hepatitis B virus infection. J Hepatol 2017;67(2):370-398.

3. Terrault NA, Lok ASF, McMahon BJ, et al. Update on prevention, diagnosis, and treatment

of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology 2018;67(4):1560-

1599.

4. Sarin SK, Kumar M, Lau GK, et al. Asian-Pacific clinical practice guidelines on the

management of hepatitis B: a 2015 update. Hepatol Int 2016;10(1):1-98.

5. Farrell GC, Wong VW, Chitturi S. NAFLD in Asia--as common and important as in the West.

Nat Rev Gastroenterol Hepatol 2013;10(5):307-318.

3

- 6. Fan JG, Kim SU, Wong VW. New trends on obesity and NAFLD in Asia. J Hepatol 2017;67(4):862-873.
- 7. Charatcharoenwitthaya P, Pongpaibul A, Kaosombatwattana U, et al. The prevalence of steatohepatitis in chronic hepatitis B patients and its impact on disease severity and treatment response. Liver Int 2017;37(4):542-551.
- 8. Mak LY, Seto WK, Hui RW, et al. Fibrosis evolution in chronic hepatitis B e antigen-negative patients across a 10-year interval. J Viral Hepat 2019;26(7):818-827.
- 9. Marcellin P, Gane E, Buti M, et al. Regression of cirrhosis during treatment with tenofovir disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up study. Lancet 2013;381(9865):468-475.
- 10. Seto WK, Fung J, Cheung KS, et al. Body-mass index is associated with fibrosis regression during long-term nucleoside analogue therapy in chronic hepatitis B. Aliment Pharmacol Ther 2016;44(10):1071-1079.
- 11. Kleiner DE, Brunt EM, Van Natta M, et al. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology 2005;41(6):1313-1321.
- 12. Brunt EM, Janney CG, Di Bisceglie AM, et al. Nonalcoholic steatohepatitis: a proposal for grading and staging the histological lesions. Am J Gastroenterol 1999;94(9):2467-2474.